CLINICAL TRIAL: NCT01386983
Title: Clinical and Economic Outcomes of Patients Utilizing Combination Therapy for Enlarged Prostates: A Henry Ford Database Assessment
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112599
Record Dates: First submitted 2011-02-28; First posted 2011-07-01 (Estimated); Results first posted 2011-07-01 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Prostatic Hyperplasia
Keywords: Enlarged prostate, 5-alpha-reductase inhibitor, alpha-blocker, acute urinary retention, surgery, early, costs; benign prostatic hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Early 5ARI Initiation: Patients with EP receiving either 5ARI monotherapy or combination therapy (AB + 5ARI) with early initiation of 5ARI (within 30 days of initiation of AB)
  Interventions: Drug: 5ARI; Drug: 5ARI + AB
- Late 5ARI Initiation: Patients with EP receiving combination therapy (AB + 5ARI) with late initiation of 5ARI (within 31 to 180 days after initiation of AB)
  Interventions: Drug: 5ARI; Drug: 5ARI + AB

INTERVENTIONS:
Drug: 5ARI — Dutasteride or Finasteride
  Other Names: Avodart® is a registered trademark of GlaxoSmithKline; Proscar® is a registered trademark of Merck
Drug: 5ARI + AB — 5ARI: Dutasteride or Finasteride AB: Doxazosin, Tamsulosin, Terazosin, or Alfuzosin
  Other Names: Proscar® is a registered trademark of Merck; Hytrin® is a registered trademark of Abbott Laboratories; Flomax® is a registered trademark of Astellas Pharma; Avodart® is a registered trademark of GlaxoSmithKline; Cardura® is a registered trademark of Pfizer Inc; Uroxatral® is a registered trademark of Sanofi-Aventis

SUMMARY:
This retrospective study aims to assess the clinical and economic impact of early initiation of 5-alpha-reductase inhibitor (5ARI) therapy in patients with enlarged prostate (EP) receiving 5ARI monotherapy or combination therapy with an alpha-blocker (AB) compared to late initiation of 5ARI therapy in patients receiving combination therapy. The Henry Ford Health System databases will be utilized for this study (2000-2008).

ELIGIBILITY:
Inclusion Criteria:

* Males
* aged 50 years or older
* medical claim of EP
* prescription claim(s) for either a 5ARI or both 5ARI and AB (provided both are within 180 days of index date)
* continuously eligible for 3 months prior to and at least 5 months after their index prescription date.

Exclusion Criteria:

* Patients with prostate or bladder cancer
* any prostate-related surgical procedure within 5 months of index date
* prescription claim for finasteride indicative of male pattern baldness; AB monotherapy only; initiation of 5ARI occurring more than 180 days after initiation of AB

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will identify eligible patient data between April 1, 2000, and December 31, 2007, and allows for patient data to be followed for 3 months prior to and up to 1 year following index prescription date.
Sampling Method: Non-Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Groups:
- Early Cohort: Participants treated either (1) only with a 5-alpha reductase inhibitor (5ARI) (monotherapy 5ARI users [dutasteride and finasteride]) (mono ARI users) or with (2) a 5ARI within 30 days of an alpha-adrenergic blocker (AB [doxazosin, tamsulosin, terazosin, and alfuzosin]) (early combination users)
- Delayed Cohort: Participants who began a 5ARI 30 days after an AB but within 180 days (late combination users)
Period: Overall Study
Arm/Group | Early Cohort | Delayed Cohort
Started | 264 | 68
Completed | 264 | 68
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Cohort | Delayed Cohort | Total
Number analyzed (Participants) | 264 | 68 | 332
Age, Customized [Number; unit: participants]
  >=50 years old | 264 | 68 | 332
  <50 years old | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 264 | 68 | 332

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Progression
Description: Participants with clinical progression are defined as those with acute urinary retention and/or receiving prostate-related surgery.
Time Frame: 3 months prior to and 12 months following index date
Population: Participants with enlarged prostate during the enrollment period (EP)/pre-index period; treated with AB and 5ARI within 180 days of index date (ID), or 5ARI only, in the EP; and with continuous Health Maintenance Organization enrollment (access to medical/pharmacy services) for at least 3 months prior to and 5 months of ID.
Measure: Number; unit: participants
Arm/Group | Early Cohort | Delayed Cohort
Number analyzed (Participants) | 264 | 68
participants | 14 | 5
Statistical Analysis 1: Comparison: Early Cohort vs Delayed Cohort; Test type: Superiority or Other; p = 0.0128, Regression, Cox; Cox Proportional Hazard = 3.406, 95% CI 2-sided [1.297 to 8.941]

2. Secondary Outcome: Dollar Amount of Enlarged Prostate (EP)-Related Medical Costs Incurred Per Month
Description: EP-related charges were defined as medical claims submitted to The Health Alliance Plan (HAP), a Health Maintenance Organization (HMO) owned and operated by the Henry Ford Heath System (HFHS) for reimbursement and internal billing data that had a primary diagnosis of EP. Charges were assessed during months 5 to 12 of the variable follow-up period. Follow-up could end only due to end of continuous eligibility, end of study period, or end of 1-year follow-up. Charges were computed on a per-month basis due to differences in the length of follow-up in the sample.
Time Frame: 3 months prior to and 12 months following index date
Population: Enrolled Population
Measure: Mean (95% Confidence Interval); unit: dollars
Arm/Group | Early Cohort | Delayed Cohort
Number analyzed (Participants) | 264 | 68
dollars | 129.14 [97.42 to 154.19] | 254.51 [178.92 to 329.41]
Statistical Analysis 1: Comparison: Early Cohort vs Delayed Cohort; Test type: Superiority or Other; p = 0.0002, Generalized linear model; Gamma distribution with log-link function was used

ADVERSE EVENTS:
Description: This was a retrospective database study, and adverse event/serious adverse event information was not captured in the study.
Arm/Group | Early Cohort | Delayed Cohort
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.